CLINICAL TRIAL: NCT02144753
Title: Use of Novel Prebiotic Fiber for Targeted Dietary Management of Irritable Bowel Syndrome (Nutrabiotix Phase II)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per DSMB, study fiber had given subjects more adverse events and made their IBS symptoms worse than the psyllium group.
Sponsor: Nutrabiotix, LLC (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SBIR-2013-NTX
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Constipation-predominant IBS (IBS-C)
Keywords: IBS-C; Constipation; IBS
MeSH Terms: conditions — Constipation | interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NTX-1 (Experimental): NTX-1 (18 g)
  Interventions: Dietary Supplement: NTX-1
- Psyllium (Active Comparator): psyllium (15 g)
  Interventions: Drug: psyllium (15 g)

INTERVENTIONS:
Dietary Supplement: NTX-1 — Investigational NTX-1 fiber to be taken as three (6g each) packets of the fiber per day, one 8g packet in the morning (one hour before eating breakfast) and the other two 8g packets in the afternoon and evening.Fasting required for the morning dose and recommended with afternoon and evening dose.
  Other Names: Nutrabiotix (18g)
  Arms: NTX-1
Drug: psyllium (15 g) — Psyllium (an over-the-counter fiber) to be taken as three (5g each) packets of the fiber per day, one 5g packet in the morning (one hour before eating breakfast) and the other two 5g packets in the afternoon and evening.Fasting required for the morning dose and recommended with afternoon and evening dose.
  Other Names: psyllium
  Arms: Psyllium

SUMMARY:
The objective of this Phase II trial is to test the NTX-1 Fiber in patients with constipation-predominant IBS (IBS-C) and determine if it can reduce symptoms, beneficially modify gut microbiota composition, and improve gut milieu in these patients. The investigators hypothesis for the Phase II study is that NTX-1 Fiber is better tolerated (i.e has less side effects) and is more effective than psyllium (the most commonly used fiber in the US) for symptom improvement and is effective in correcting the abnormal colonic milieu in those with dysbiosis and low SCFA levels.

DETAILED DESCRIPTION:
The investigators will conduct an 18-week (2-week initial run-in phase, 12-week treatment phase, and 4-week follow up phase), 2-arm, randomized, double-blind, controlled Phase 2 trial in 120 subjects with IBS-C. A 2-week run in will be completed in order to ensure the stability of baseline symptom scores and to ensure that all study subjects have the required symptom severity to fulfill the inclusion criteria before randomization and beginning the treatment. The investigators selected a 12-week treatment phase because of the adequacy of this length of time to clinically see the impact of fiber supplementation (as seen in the investigators Phase I trial), and because of the 12-week duration requirement of the FDA for all therapeutic intervention/agents for treatment of IBS. The 4-week follow up phase is to determine the sustainability of the effects of therapy and to obtain further safety data.Potential study subjects will be identified though the Rush University Medical Center (RUMC) clinical databases; advertisements on the RUMC clinical trials and GI websites, RUMC Facebook and other social media sites; and IRB approved flyers placed in the GI clinic and throughout the medical center. All potential candidates will be interviewed on the phone by a clinical coordinator using a structured checklist, at which time the study requirements will also be explained. Subjects will be asked for food allergies, including artificial sweeteners such as sucralose and ascelfame K. Subjects will also be informed that the fiber is made out of corn or psyllium and not other grains. However, it can't be guaranteed that it is free of other food allergy-related contaminants. Also, subjects will be asked to limit intake of foods containing more than 3 grams of prebiotics. A list of these foods will be provided.

Those who are eligible and are willing to participate will be invited for the first study visit. Five visits will be required from each subject.

Visit 1: After the subject has reviewed and signed the informed consent form, the investigators will check to see if they are eligible for this study by a physical exam, questionnaires and a blood test. A physician or their assistant will do a physical exam and take the subjects vitals (such as height, weight, waist circumference and blood pressure).

The Subject Information Form will be an administered questionnaire related to their health, disease, and their family medical history. They will then have 2½ tablespoons of blood drawn by a certified nurse or medical assistant. They will be reminded in advance to fast 12 hours prior to their research visit. The blood tests include: CBC, CMP, CRP, TSH, INR, fasting lipid profile and HbA1c. The subject will be given a 3-day food diary and a 14-day IBS symptom diary to complete before their next visit. They will also be provided with stool collection supplies and instructions to take home. When blood test results are available, those who do not fit the criteria will be called within 7 days after Visit 1 stating that they are ineligible. Among these blood tests, the fasting lipid profile results will be given to the subject after their participation in the study and after completion of the study. The rest of the results will be given to the subject at their next visit. If they continue to be a candidate in this study based on blood results, the potential subjects will fill out the 3-day food diary, continue to fill out the 14-day IBS symptom diary, and complete the stool collection the day before or the morning of Visit 2. The subject will be advised to not keep the stool at room temperature longer than 5 hours. If they anticipate it to be longer than 5 hours before their visit time, then the stool will be kept in the freezer. Both of the diaries and the stool sample are to be brought to Visit 2, which is 2 weeks after their Visit 1. Visit 1 will be about 3 hours in length.

Visit 2: The subject will give the study coordinator their 3-day food diary, 14-day IBS symptom diary, and stool sample. They will provide the date of stool collection, as well as the method of storing the sample. The physician will review their 14-day IBS symptom diary and confirm their eligibility. If they continue to be eligible, the physician will do a physical exam and take their vitals (such as weight, waist circumference and blood pressure). The subject will then be asked to fill out a series of questionnaires relating to their diet (VioScreen Food Frequency Questionnaire), IBS symptoms (IBS-Quality of Life questionnaire [IBS-QoL] and IBS Questionnaire by Whorwell and Francis), sleeping/circadian patterns (2 NIH sleep questionnaires, Munich Chronotype Questionnaire, Lark/Hummingbird/Owl questionnaire, food timing questionnaire), the Expectancy and Credibility Questionnaire, and the 34-item tool asking about their GI symptoms and severity. The subject will then be randomized into one of the two groups. Depending on which group they are randomized to, they will be provided with a 6-week supply of NTX-1 OR psyllium fiber products in an identical appearing sachet along with instructions for taking the fiber. They will be provided with a 3-day food diary and a daily and weekly IBS symptom diary to fill out prior to Visit 3. This visit will be about 3 hours in length. The next visit will be 6 weeks after Visit 2.

Visit 3: The subject will give the study coordinator their 3-day food diary, the daily and weekly IBS symptom diary, and any excess fiber product. The physician will review their IBS symptom diary and ensure there are no significant adverse events. The physician will do a physical exam and take their vitals (such as weight, waist circumference and blood pressure). The subject will then be asked to fill out a series of questionnaires relating to their IBS symptoms (IBS-Quality of Life questionnaire (IBS-QoL) and IBS Questionnaire by Whorwell and Francis), sleeping/circadian patterns (2 NIH sleep questionnaires, Munich Chronotype Questionnaire, Lark/Hummingbird/Owl questionnaire, food timing questionnaire), the Expectancy and Credibility Questionnaire, and the 34-item tool asking about their GI symptoms and severity. Next, they will have 2 tablespoons of blood drawn by a certified nurse or medical assistant. The following blood tests will be done: CBC, CMP and CRP. The subject will be reminded in advance to fast 12 hours prior to their research visit. A copy of their blood test results will be given to them at their next visit. Next, they will be given another 6-week supply of the fiber product, the 3-day food diary, a daily and weekly IBS symptom diary to fill out prior to Visit 4 and stool collection supplies. They are asked to collect stool as previously indicated and bring the stool to Visit 4; handling will be identical to previous visit. This visit will be about 2 hours in length. The next visit will be 6 weeks after their Visit 3.

Visit 4: The subject will give the study coordinator their 3-day food diary, the daily and weekly IBS symptom diary, and any excess fiber product. The physician will review their IBS symptom diary and ensure there are no significant adverse events. The physician will complete a physical exam and take their vitals (such as weight, waist circumference and blood pressure). The subject will then be asked to fill out a series of questionnaires relating to their diet (VioScreen Food Frequency Questionnaire), IBS symptoms (IBS-Quality of Life questionnaire (IBS-QoL) and IBS Questionnaire by Whorwell and Francis), sleeping/circadian patterns (2 NIH sleep questionnaires, Munich Chronotype Questionnaire, Lark/Hummingbird/Owl questionnaire, food timing questionnaire), the Expectancy and Credibility Questionnaire, and the 34-item tool asking about their GI symptoms and severity. They will then have 2½ tablespoons of blood drawn by a certified nurse or medical assistant. Subjects will be reminded in advance to fast 12 hours prior to their research visit. The blood tests include: CBC, CMP, CRP, TSH, INR, fasting lipid profile and HbA1c. Among these blood tests, the fasting lipid profile results will be given to the subject after the completion of the study. The rest of the results will be given to the subject at their next visit. They will be provided with a 3-day food diary and a daily and weekly IBS symptom diary to fill out prior to Visit 5. Visit 4 will be about 3 hours in length. The next visit will be 4 weeks after their fourth visit, which is the subjects' last visit.

Visit 5: The subject will give the study coordinator their 3-day food diary and the daily and weekly IBS symptom diary. The physician will review their IBS symptom diary and ensure there are no significant adverse events. The physician will do a physical exam and take their vitals (such as weight, waist circumference and blood pressure). The subject will then be asked to fill out questionnaires relating to their IBS symptoms (IBS-Quality of Life questionnaire (IBS-QoL) and IBS Questionnaire by Whorwell and Francis) and the 34-item tool asking about their GI symptoms and severity. Next, they will have 2 tablespoons of blood drawn by a certified nurse or medical assistant. Subjects will have been reminded in advance to fast 12 hours prior to their research visit. The following blood tests will be done: CBC and CMP. A copy of their blood test results, including the two fasting lipid profile tests, will be given to the subject via e-mail or mail. This visit will be about 2 hours in length.

ELIGIBILITY:
Inclusion - History

1. Between the ages of 18-75
2. Have recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months
3. Have at least 2 of the following in the last 6 months:

   1. Improvement of abdominal pain or discomfort with defecation
   2. Onset of abdominal pain or discomfort associated with change in frequency of stool
   3. Onset of abdominal pain or discomfort associated with a change in form/appearance of stool
4. Symptom onset at least 6 months prior to screening date
5. Willing to take study supplement three times a day and willing to comply with all study procedures (i.e. swallow capsules)
6. Willing to stop taking over-the-counter laxatives after the 2 week screening period (Ex: ex-lax, senna, miralax, milk of magnesia)

   Inclusion - Screening Diary
7. Abdominal bloating/discomfort/pain (if either a, b, OR c is positive, then this meets the criteria for #7)

   1. A weekly average of worst abdominal bloating score of ≥ 3 during the screening period on a 0-10 numeric rating scale
   2. A weekly average of worst abdominal discomfort score of ≥ 3 during the screening period on a 0-10 numeric rating scale
   3. A weekly average of worst abdominal pain score of ≥ 3 during the screening period on a 0-10 numeric rating scale
8. Bowel movements/stool consistency (if either a OR b is positive, then this meets the criteria for #8)

   1. Less than 3 spontaneous complete BM (SCBM) per week. (SCBM is defined as a BM occurring in the absence of a laxative that is associated with a sense of complete evacuation)
   2. Stool consistency of 1-2 on Bristol scale at least twice a week OR >25% of BM for the week

Exclusion- Lab Results

1. Abnormalities in CBC (Hgb<12 g/dL, platelet count<100000, WBC<4000 or >10000)
2. Abnormal liver function tests (ALT, AST, alkaline phosphatase, or bilirubin >1.5 times normal range)
3. Abnormal renal function tests (BUN or creatinine >1.5 times normal range)
4. Low serum albumin (<3 g/dL)
5. Uncontrolled thyroid disease as evident from abnormal TSH level
6. High CRP (> 5), except those evaluated for IBD and IBD is ruled out through colonoscopy, CT or additional tests
7. Insulin-requiring and/or poorly controlled diabetes (well-controlled diabetics with HbA1c <7 may be enrolled)

   Exclusion- History
8. Patient history of GI diseases (except for hemorrhoids or occasional (<3 times a week) heartburn)

   1. Inflammatory bowel disease (Ex: ulcerative colitis, crohn's disease, any colitis)
   2. Celiac disease
   3. Colonic inertia (lazy/slow colon resulting in surgery, resection or daily laxatives)
   4. Diverticular stricture (narrowing of the colon)
9. Antibiotic use within last 4 weeks
10. Severe uncontrolled hypertension
11. Significant uncompensated cardiac or respiratory diseases (defined as requiring daily medication for management of their diseases (Ex: on oxygen or can't walk))
12. Prior extensive intestinal resection
13. History of psychiatric hospitalization OR suicide attempt in the last 5 years
14. Drug and/or alcohol abuse
15. Plan to have a major change of their dietary habit during the following 5 months
16. Drug induced constipation (Ex: opiates)
17. Pregnant or lactating
18. Use of narcotic medications (pain killers, Ex: hydrocodone, methadone, morphine, oxycodone or tramadol) or anticoagulant/antiplatelet agents (ex: heparin, warfarin , dabigitran., Coumadin)
19. If the subject is older than 50 years of age, subjects who have not had a colonoscopy within last 7 years or CT colonography within last 5 years to rule out colon cancer
20. Alarm symptoms of colon cancer such as:

    1. Weight loss (>10% unintentional loss of body weight in last 6 months)
    2. Blood in the stool (except for clearly documented hemorrhoidal bleed OR colonoscopy excluding colon cancer within the last year for blood in the stool)
    3. Anemia (without a full work-up, including a colonoscopy or other tests deemed important)
21. Continued chronic and daily use of prescription laxatives (Ex: Amitiza or Linzess/ linaclotide in the last month)
22. Loose or watery stools > than 3 times per week
23. History of fecal impaction requiring disimpaction in the last 3 months
24. History of laxative abuse (Ex: eating disorders)
25. Use of medications that affect gastrointestinal motility (i.e. resolor, domperidone, reglan, cisapride, anticolonergic drugs, tricyclic antidepressant [Ex: Amitriptyline, Amoxapine, anafranil, asendin, elavil, norpramin/desipramine, doxepin, pamelor/nortriptyline, sinequan, surmontil/trimipramine, tofranil/imipramine or vivactil/protriptyline]) SSRI's are OK
26. Documented untreated pelvic floor dysfunction
27. Colonic organic diseases such as:

    1. Current colonic cancer or strictures
    2. Connective tissue disease (ex: scleroderma, lupus)
    3. Other neurological disorders leading to chronic constipation (Ex: Parkinson's or multiple sclerosis)
28. Dietary intake exceptionally high in plant-based, high fiber foods, including those following a strict vegetarian diet (high fiber foods: fruits, vegetables, beans, whole grains, fortified foods)
29. Consumption of probiotics, prebiotics, or synbiotics without an appropriate 2-week washout period (Ex: Activia, FiberOne products, probiotics supplements such as Align, Pearls, or fiber/prebiotic supplements such as Metamucil, Benefiber, Citrucel, Fiber Choice, Fiber Powder)
30. Intention of using fiber products during the study (other than the study supplement)
31. Known food allergies or hypersensitivities (Ex: the components of psyllium or NTX-1 (corn))
32. Have a colonoscopy done within the next 5 months

Exclusion- Screening Diary 32. Use of laxatives more than twice in the screening period (The following are the ONLY laxatives the subject is allowed to use during the screening period: Ex-lax, senna, miralax and milk of magnesia) 33. Have not completed 11 out of 14 days of symptoms diary at screening 34. Have an average daily IBS-C global symptom score of <2 in the screening period 35. Average Bristol stool scale of more than 4 within the screening period 36. Loose or watery stools with Bristol stool scale of 5 or greater for a total of 6 or more days during the screening period 37. Use of fiber products during the screening period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Composite improvement in the following three areas: IBS global improvement score on the Likert Scale, frequency & consistency of stools, & severity of abdominal pain, discomfort and bloating | up to 14 months
  Compare the effects of NTX-1 (18 grams) against psyllium (15 grams) on IBS global improvement score, frequency & consistency of stools, & severity of abdominal pain, discomfort and bloating in patients with IBS-C (as defined by the Rome III criteria).

SECONDARY OUTCOMES:
Determine side effects of NTX-1 | up to 14 months
  The following scales will be used to measure side effects experienced by subjects: (1) Frequency (# of total BM/week) and consistency of stool (Bristol stool scale); (2) Severity of abdominal pain (11 point numeric scale from 0-10); (3) Severity of bloating (11 point numeric scale from 0-10); (4) Severity of abdominal discomfort (11 point numeric scale from 0-10); (5) Difficulty with defecation (i.e. straining) (11 point numeric scale from 0-10); (6) Frequency (number of SCBMs/week and SBMs/week), (7) Global IBS symptom score from 0-4 on a 5 point numeric scale/week; (8) Adequate relief from IBS symptoms (yes, no)

CONTACTS AND LOCATIONS:
Overall Officials: Ece Mutlu, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States